CLINICAL TRIAL: NCT02469493
Title: The Effect and Mechanism of Electroacupuncture on Acute Chemotherapy-induced Nausea and Vomiting
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xidian University (Other)
Responsible Party: Principal Investigator, Wei Qin, Professor, Xidian University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2014CB543203
Record Dates: First submitted 2015-06-08; First posted 2015-06-11 (Estimated); Last update posted 2015-06-22 (Estimated); Status verified 2015-06

CONDITIONS: Lung Neoplasms
MeSH Terms: conditions — Lung Neoplasms | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Acupuncture 1 (Experimental): In this group, patients separately received twice electroacupuncture at bilateral PC6 acupoint before and after Cisplatin administration on the first day of chemotherapy.
  Interventions: Device: acupuncture (Huatuo)
- Acupuncture 2 (Experimental): In this group, patients separately received twice electroacupuncture at bilateral PC6 and RN12 acupoints before and after Cisplatin administration on the first day of chemotherapy.
  Interventions: Device: acupuncture (Huatuo)
- Sham acupuncture (Sham Comparator): In this group, patients separately received twice electroacupuncture at bilateral nonacupuncture point (S1 located at lateral of flexor carpi radialis, 2 cun above the wrist. S2 located at 3 cun right side of RN12) before and after Cisplatin administration on the first day of chemotherapy.
  Interventions: Device: acupuncture (Huatuo)
- Waitinglist control (No Intervention): In this group, patients received no electroacupuncture

INTERVENTIONS:
Device: acupuncture (Huatuo) — The needles used were Huatuo brand (Suzhou, China) sterile disposable stainless steel filiform; needles sized 0.25*25 mm. After disinfection, needles were inserted 0.5 to 0.8 inches into the skin and were manipulated manually to obtain Deqi. An electric stimulator (Huatuo SDZ-V, Suzhou, China) was connected to the needles and delivered a constant-current, 0.2-ms, density-wave, stimulus of 2 to 10-Hz frequency, level of intensity was as much as tolerable, but not painful to the subjects. The needles were left for 30 minutes and then removed.
  Arms: Acupuncture 1; Acupuncture 2; Sham acupuncture

SUMMARY:
The purpose of this study is to compare the preventive effect of electroacupuncture and sham acupuncture on acute chemotherapy-induced nausea and vomiting and then investigate its potential mechanism by using functional Magnetic Resonance Imaging (fMRI).

ELIGIBILITY:
Inclusion Criteria:

* First diagnosed stage Ⅲ-Ⅳ lung cancer patients on cisplatin chemotherapy;
* Right-handed and aged 18 to 75 years;
* Karnosky performance status (KPS) ≥ 70;
* Life expectancy ≥ 6 months.

Exclusion Criteria:

* Had brain metastases or other concurrent life-threatening diseases;
* Nausea and/or vomiting were present 24h before chemotherapy treatment;
* Suffered from or had a history of gastrointestinal diseases;
* Had a history of head trauma, serious neurological or psychiatric disorders;
* Participating in other clinical trials currently;
* Had any contraindication to exposure to a high magnetic field or receive acupuncture

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2015-01; Primary Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
The scores of Rhodes Index of Nausea, Vomiting and Retching. | 24 hours

SECONDARY OUTCOMES:
Content of 5-hiaa in urine | 12 hours
Heart Rate Variability | 1 hour
Tachygastria percentage | 1 hour
Dosage of antiemetic drugs | 24 hours

OTHER OUTCOMES:
Neuroimaging data | 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Xijing Hospital, Xi'an, Shaanxi, China